CLINICAL TRIAL: NCT02367638
Title: A Single-center, Dose Block-randomized, Single-blind, Active-controlled, Dose Escalation Phase 1 Clinical Trial to Evaluate the Safety and Efficacy (Immunogenicity) of MG1111 in Healthy Adults
Brief Title: Dose-escalation Phase 1 to Evaluate the Safety and Efficacy of MG1111 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MG1111_P1
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Varicella (Chicken Pox)
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MG1111 (Experimental)
  Interventions: Biological: MG1111
- VARIVAX (Active Comparator)
  Interventions: Biological: VARIVAX

INTERVENTIONS:
Biological: MG1111 — Low, Medium, High Plaque-Forming Unit (PFU) of MG1111 in 0.5 mL dose is administered by subcutaneous injection
  Arms: MG1111
Biological: VARIVAX — VARIVAX is administered by subcutaneous injection
  Arms: VARIVAX

SUMMARY:
The purpose of this study is to determine whether varicella live vaccine is safe and effective in the healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female individuals between 20 and 55 years of age at screening test

   * In the case of female, individuals must be applicable for one of the following;
   * In the case of female of childbearing potential, any negative pregnancy test using urine hCG at screening
   * Menopausal for at least 2 years
   * Surgical sterilization (status after hysterectomy, bilateral oophorectomy, bilateral tubal ligation or the status using other contraceptive methods)
   * Monogamous relationship with vasectomized partner prior to screening visit
   * Individuals who are used acceptable contraceptive methods from 3 month prior to the subject's study entry to 1 month after vaccination (acceptable contraceptive methods; condom, diaphragm or cervical cap)
2. If male who is sexually active with the female "of childbearing potential" , the individuals who agree to use any of the acceptable contraceptive methods during this study period and agree to not donate the sperm until 1 month
3. At screening visits, individuals who are over 55 kg in man, over 50kg in woman and whose ideal body weight is within 20 % ((ideal body weight = (height -100)*0.9)
4. Individual who has no clinically significant abnormalities in screening test within 28 days prior to vaccination
5. Individuals who were voluntarily signed informed consent form after receiving education about this study and able to comply with the requirements for the study

Exclusion Criteria:

1. Individuals who received any other vaccines within 4 weeks prior to the screening visit
2. Individuals who are planning to receive the other vaccines during this study
3. Individuals who had wound, scar, tattoo, dermatological disorders or injection affecting safety evaluation
4. Individuals with alcohol or caffeine abuse or heavy smoker (caffeine : >5 cups/day, alcohol : 210g/week, smoke : 10 /day)
5. Individuals who received any other investigational product within 90 days prior to vaccination
6. individuals who donated the whole blood within 60 days or apheresis within 30 days prior to vaccinating investigational product
7. Individuals who administered with another prescription medicine, herbal medicine within 14 days or over-the-counter drug or vitamins within 7 days before vaccination
8. Individuals with history or illness affecting immune system (1) individuals with continuously anti-viral therapy within 6 months prior to participating in this study (2) Individuals with leukemia, lymphoma, other malignant neoplasm or hematodyscrasia affecting the bone marrow or lymphatic system (3) Immunodeficient individuals (primary or acquired immunodeficiency states, immunodeficiency, hypogammaglobulinemia, dysgammaglobulinemia) (4) Individuals who are receiving immunosuppressive therapy (5) Individuals who have treated immunoglobulin or blood-derived products within 6 months of enrollment (6) Individuals with a family history of congenital or hereditary immunodeficiency
9. Individuals with any clinically relevant history of other disease or disorder - gastrointestinal, respiratory, renal, hepatic, neurological (Guillain-Barre syndrome), psychiatric or malignant tumor
10. Individuals with any febrile illness or body temperature ≥38℃ before vaccination
11. Individuals known hypersensitivity or allergy to components of investigational product (including gelatin and neomycin)
12. Individuals who are any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG, and clinical laboratory tests
13. Pregnancy or breastfeeding
14. Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the solicited adverse events and unsolicited adverse events during 7 days after vaccination | 7 days
To evaluate the unsolicited adverse events during 42 days after vaccination | 42 days

SECONDARY OUTCOMES:
To evaluate the efficacy of Geometric mean titer (GMT) and GMT ratio using FAMA assay antibody titer at Day 42 | 42 days
To evaluate the efficacy of Geometric mean titer (GMT) and GMT ratio using gpELISA antibody titer at Day 42 | 42 days